CLINICAL TRIAL: NCT06953986
Title: Study Comparing Vonaprazan 10 mg, Vonaprazan 20 mg, and Esomeprazole 40 mg for the Healing of LA Grade B or Higher Reflux Esophagitis at 8 Weeks
Brief Title: A Randomized, Three-Arm Study Comparing Vonaprazan 10 mg, Vonaprazan 20 mg, and Esomeprazole 40 mg for the Healing of LA Grade B or Higher Reflux Esophagitis at 8 Weeks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: VNP2025
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- To determine whether Vonaprazon 10mg heals grade B esophagitis at 8 weeks (Other): Vonaprazon 10 mg heals gerd symptoms after 8 weeks
  Interventions: Drug: Vonoprazan
- To determine whether Vonaprazon 20mg heals grade B esophagitis at 8 weeks (Other): Vonaprazon 20 mg heals gerd symptoms after 8 weeks
  Interventions: Drug: Vonoprazan
- To determine whether esomeprazole 40mg heals grade B esophagitis at 8 weeks (Other): Esomeprazole 40mg heals gerd symptoms after 8 weeks
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: Vonoprazan — Vonaprazon is potassium competitive acid blockers
  Other Names: PCAB
  Arms: To determine whether Vonaprazon 10mg heals grade B esophagitis at 8 weeks; To determine whether Vonaprazon 20mg heals grade B esophagitis at 8 weeks
Drug: Esomeprazole 40mg — esomeprazole is a proton pump inhibitor as it prevents excess of gastric acid secretion in the stomach
  Other Names: Proton pump inhibitor
  Arms: To determine whether esomeprazole 40mg heals grade B esophagitis at 8 weeks

SUMMARY:
Primary Objective

• To compare the healing rates of LA grade B or higher reflux esophagitis at 8 weeks among patients treated with Vonaprazan 10 mg, Vonaprazan 20 mg, and Esomeprazole 40 mg once daily.

Secondary Objectives

* To assess the improvement in reflux symptoms using the GERD-Q score at 8 weeks.
* To evaluate the incidence of adverse events across treatment groups.

DETAILED DESCRIPTION:
Study Design:

* This is a randomized, open-label, parallel-group, non-inferiority trial. Randomization and Blinding
* Participants will be randomized in a 1:1:1 ratio to receive Vonaprazan 10 mg, Vonaprazan 20 mg, or Esomeprazole 40 mg once daily for 8 weeks.
* Randomization will be stratified by baseline severity of esophagitis (LA grade B vs. C/D).
* The study will be open-label, but the outcome assessors will be blinded. Study Arms

  1. Vonaprazan 10 mg once daily
  2. Vonaprazan 20 mg once daily
  3. Esomeprazole 40 mg once daily

     Duration:
* 8 weeks of treatment, followed by endoscopic assessment and symptom evaluation.

I

Study Procedures:

Baseline :

* Perform upper GI endoscopy to confirm LA grade B or higher esophagitis.
* Record baseline GERD-Q score.
* Randomize participants into one of the three treatment groups.
* Dispense study medication. Follow-up (Week 4 - Interim Assessment)
* Assess GERD-Q score.
* Monitor adherence and adverse events. End-of-Treatment (Week 8 - Primary Outcome Assessment)
* Repeat upper GI endoscopy to assess mucosal healing.
* Reassess GERD-Q score.
* Collect adverse event data.
* Conclude study participation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Endoscopically confirmed LA grade B, C, or D reflux esophagitis.
* GERD symptoms (heartburn, regurgitation) for at least 4 weeks prior to enrollment.
* Willing to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Previous or ongoing treatment with Vonaprazan or Esomeprazole in the last 4 weeks.
* Prior esophageal surgery or radiation therapy.
* Barrett's esophagus, esophageal stricture, or malignancy.
* Pregnant or breastfeeding women.
* History of PPI-refractory GERD or severe gastroparesis.
* Significant hepatic or renal impairment (ALT/AST >3× ULN, eGFR <30 mL/min).
* Use of NSAIDs, steroids, or anticoagulants affecting healing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2025-06-07 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
• Endoscopic healing of reflux esophagitis at 8 weeks (defined as resolution of LA grade B, C, or D esophagitis). | 8 weeks
  healing of ulcers after taking vonaprazon 10mg, 20 mg
Endoscopic healing of reflux esophagitis at 8 weeks (defined as resolution of LA grade B, C, or D esophagitis). | 8 weeks
  healing of ulcers after taking esomeprazole 40mg

SECONDARY OUTCOMES:
• GERD-Q score improvement at 8 weeks (compared to baseline). | 8 weeks
  symtoms improvement like heartburn, regurgitation which can be calculated with scale 1 (mild symptoms ) to 5 (worse symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MD DM, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology /Aig Hospitals, Hyderabad, Telangana, India